CLINICAL TRIAL: NCT00304356
Title: Compassionate Use of Nitazoxanide for the Treatment of Clostridium Difficile Colitis in Patients Who Have Failed Conventional Therapy
Brief Title: Compassionate Use of Nitazoxanide for the Treatment of Clostridium Difficile Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daniel M. Musher MD (U.S. Federal Agency)
Collaborators: Baylor College of Medicine (Other)
Responsible Party: Sponsor-Investigator, Daniel M. Musher MD, PI, Michael E. DeBakey VA Medical Center
Organization: Michael E. DeBakey VA Medical Center (U.S. Federal Agency)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-15601
Record Dates: First submitted 2006-03-16; First posted 2006-03-17 (Estimated); Results first posted 2017-12-15 (Actual); Last update posted 2017-12-15 (Actual); Status verified 2017-05

CONDITIONS: Clostridium Enterocolitis; Pseudomembranous Colitis
Keywords: Clostridium difficile Associated Diarrhea
MeSH Terms: conditions — Enterocolitis, Pseudomembranous | interventions — nitazoxanide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- active drug (Other): 500 mg nitazoxanide bid given to patient
  Interventions: Drug: Nitazoxanide

INTERVENTIONS:
Drug: Nitazoxanide — 500 mg bid
  Other Names: alinia

SUMMARY:
The purpose of this study is for compassionate use of nitazoxanide in the treatment of diarrheal disease due to Clostridium difficile infection when the patient has failed previous treatment with metronidazole or vancomycin.

DETAILED DESCRIPTION:
Clostridium difficile is the leading cause of nosocomial diarrheal disease associated with antibiotic therapy. This is a debilitating condition with substantial morbidity and a mortality that may be around 2-3%. There has been an enormous increase in this disease at the VA Medical Center during the past two years, just as has occurred at other hospitals throughout the United States.

Currently recommended therapy for this condition is metronidazole, given orally. About 15-20% of patients fail to respond to initial therapy with metronidazole, and another 20% relapse after treatment. Relapses may be treated with another course of metronidazole; about one-half will respond to this therapy. The failures are treated with oral vancomycin, but this drug also has a failure rate of 10-20%. There is, at present, no other accepted therapy (although some articles in the literature favor vancomycin with ingested bacteria from benign species). Furthermore, there is a strong risk to the emergence of resistant bacteria when hospitalized patients are treated with oral vancomycin.

Nitazoxanide is an FDA approved drug that is marketed in the U.S. and has been widely used throughout the world to treat parasitic diseases of the gastrointestinal tract; several million children have been treated with this drug during the past decade. Nitazoxanide has been approved as an antiprotozoal agent for oral administration in pediatric patients, ages 1 through 11, with diarrhea. The drug acts by interfering with anaerobic metabolic pathways, and it has been shown to have excellent in vitro activity against C. difficile. We hypothesized that this drug was both safe and effective as an alternative in patients who have diarrheal disease caused by C. difficile. The IRB approved a double-blind protocol to compare metronidazole with nitazoxanide, and we have treated a total of 16 patients so far under this protocol.

In our IRB-approved double blind study (by design, two thirds of the subjects have been randomized to the nitazoxanide), our patients have appeared to have a good response rate -- so good, in fact, that we think that nitazoxanide may be a better drug to treat this infection than either metronidazole or vancomycin.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be > 18 years of age
* Clinical diagnosis of C. difficile associated disease, based on the new onset of diarrhea, abdominal discomfort, or otherwise unexplained fever or leukocytosis
* Diagnosis of C. difficile colitis proven by positive assay for C. difficile toxin in feces
* Disease has been treated, and the symptoms failed to respond to treatment with metronidazole or vancomycin, or symptoms promptly relapsed after completing a course of therapy with either of these drugs
* Able to take oral medication

Exclusion Criteria:

* Patients with other recognized causes of diarrhea or colitis
* Women of child bearing age who are pregnant, breast feeding, or not using birth control
* Patients taking coumadin, phenytoin, celecoxib, or losartan
* Patients with renal insufficiency (BUN or creatinine >2 times baseline)
* Serious systemic disorder incompatible with the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2004-01; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M Musher, M.D., Principal Investigator — Baylor College of Medicine, Houston VA Medical Center
Locations (2):
- United States (2):
  - Baylor College of Medicine, Houston, Texas
  - Michael E. Debakey VA Medical Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Chart review at the Houston VA for patients treated with Nitazoxanide who have failed previous therapy.
Pre-assignment Details: This is a retrospective chart review.
Period: Nitazoxanide
Arm/Group | Nitazoxanide
Started | 27
Completed | 22
Not Completed | 5
Not completed — Physician Decision | 5
Period: Nitazoxanide
Arm/Group | Nitazoxanide
Started | 27
Completed | 22
Not Completed | 5
Not completed — Physician Decision | 1
Not completed — number is 0 | 1
Not completed — Physician Decision | 1
Not completed — Physician Decision | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Groups:
- Nitazoxanide: Patients with C. difficle who exhibit diarrhea and received nitazoxanide.
Arm/Group | Nitazoxanide
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27 (27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 27
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Nitazoxanide
Description: stopping of diarrhea
Time Frame: 30 days
Measure: Number; unit: participants
Groups:
- Nitazoxanide: time diarrhea from C. difficile stopped.
Arm/Group | Nitazoxanide
Number analyzed (Participants) | 27
participants | 27

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Nitazoxanide
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No